CLINICAL TRIAL: NCT06347315
Title: COGNIKET-MCI Trial: A Prospective, Randomized, Double-blind, Placebo-controlled, Multi-center, Multi-country, Pivotal Trial to Study the Effects of a Nutritional Intervention of Ketogenic Medium-chain Triglycerides (kMCT) and B-vitamins on Cognitive Functioning in Older Adults With Mild Cognitive Impairment
Brief Title: Evaluation of the Effects of a Nutritional Intervention of Ketogenic Medium-chain Triglycerides and B-vitamins on Cognitive Functioning in Older Adults With Mild Cognitive Impairment (COGNIKET-MCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2302.CLI
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: parallel and pivotal
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BrainXpert (Active Comparator): 15 g kMCT + B-vitamins (B3, B6, B9/folic acid, and B12) will be provided in powder format
  Interventions: Dietary Supplement: BrainXpert
- Placebo (Placebo Comparator): high-oleic acid sunflower oil as a calorie-equivalent, non-ketogenic vegetable oil, non added vitamin product will be provided in a powder format
  .
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: BrainXpert — sachet/stickpack of 25 g, has no preservatives, no flavors, no sweeteners, and no colorants.
  Arms: BrainXpert
Other: Placebo — high-oleic acid sunflower oil as a calorie-equivalent, non-ketogenic vegetable oil, non added vitamin product will also be provided in a powder format in a sachet/stickpack of 25 g.
  Arms: Placebo

SUMMARY:
Evaluation of the Effects of a Nutritional Intervention of Ketogenic Medium-chain Triglycerides and B-vitamins on Cognitive Functioning in Older Adults With Mild Cognitive Impairment (COGNIKET-MCI)

ELIGIBILITY:
Inclusion Criteria:

1. Have read, understood, and signed the informed consent form (ICF).
2. Be aged ≥60 years at the time of screening.
3. Presence of acquired memory complaints with a duration of >3 months. Here we refer to memory/cognitive complaints in a broader sense that can involve other cognitive domains other than memory. (As reported by the participant or reliable trial informant. Trial informants can be a relative, spouse or domestic partner, or close friend who interacts closely enough with the participant to be able to respond to assessments/questionnaires as needed.)
4. Have a clinical diagnosis of MCI (with a clinical phenotype compatible with AD, insidious SVD [ie, no post-stroke cognitive impairment], or mixed AD/SVD) according to the participating site, or referring center, aligned with international/national standards for MCI diagnosis, and additionally informed by a minimum of one of the following objective criteria as assessed by components of the Consortium to Establish a Registry for Alzheimer's Disease neuropsychological battery (CERAD NB):

   1. Word list memory task: ≤19,
   2. Word list recall: ≤5,
   3. Fifteen-item subset of the Boston Naming Test (BNT): ≤13,
   4. Constructional praxis recall: ≤7, or
   5. Total CERAD score: ≤70.
5. Full autonomy for daily living based on the Instrumental Activities of Daily Living (IADL)-Lawton scale:

   1. Score for women: 8 or
   2. Score for men: 5.
6. Participants must have an available trial informant willing and able to attend the following 3 clinic visits with the participant: V1/randomization, V3/12-month visit, and V4/18-month visit.
7. Participants must have a trial informant who in the opinion of the investigator, has contact with the trial participant for a sufficient number of hours per week (at least 2 hours per day and a minimum of 4 times per week).
8. Participants and their trial informants have an adequate ability to read and write, as well as adequate vision and hearing for neuropsychological testing according to the investigator's judgment (corrective aids are allowed).
9. CDR global score of 0 to 0.5 at screening.
10. Sexually active females of childbearing potential (defined in further detail in Appendix 1 of the protocol) must practice 2 different highly effective methods of contraception with their heterosexual partner or remain abstinent during the trial and for 30 days after the last dose of nutritional formulation. If employing contraception, the highly effective methods of contraception detailed in Appendix 1 of the protocol must be followed.
11. Females of childbearing potential must have a negative highly sensitive urine pregnancy test before randomization; a positive urine pregnancy test result must immediately be confirmed using a serum test.
12. Participants able to satisfactorily comply with the protocol requirements.
13. Participants willing and able to discontinue all prohibited concomitant medications to meet any protocol-required washout periods before and during the trial period (Section 9.6.1 of the protocol provides more details).

Exclusion Criteria:

1. Diagnosis of a major neurocognitive disorder according to the 5th Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), or dementia according to the DSM-IV and the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimer's Disease and Related Disorders Association criteria at the time of enrollment.
2. MCI related to past or recent concussion, COVID-19, or other specific etiologies (including neurodegenerative disease like Parkinson's disease, multiple sclerosis, Huntington's disease, Lewy-body disease, fronto temporal dementia), or associated with medication/substance use, per the investigator's judgment.
3. A history of COVID-19 ≤120 days before screening or completion of a vaccination course against severe acute respiratory syndrome coronavirus 2 ≤14 days before screening. The vaccine received must have been authorized for emergency use or approved by the US Food and Drug Administration.
4. Newly introduced, or change in dose, within the last 2 months before randomization, of physician-prescribed interventions or medications affecting cognition or AD (eg, acetylcholinesterase inhibitors, memantine, anti-amyloid-beta agents), or planned introduction of such medications during the trial.
5. Participants who will likely require prohibited concomitant therapy during the trial based on the investigator's judgment.
6. Known history of or ongoing alcohol or substance use disorder, based on medical history, that in the opinion of the investigator may conflict with the participant's participation.
7. Participants who, in the opinion of the investigator, medical monitor, or sponsor should not participate in the trial.
8. Symptoms suggestive of depression or anxiety according to the Hospital Anxiety and Depression Scale (HADS):

   1. HADS-D ≥8 or
   2. HADS-A ≥8.
9. Known active HIV infection, COVID, hepatitis B, or hepatitis C based on medical history.
10. Participants with epilepsy or a history of seizures, except for a single childhood febrile seizure, post-traumatic seizure, or alcohol withdrawal seizure.
11. Participants considered to be in poor general health based on the investigator's judgment. Examples include participants who have recent clinically significant weight loss, chronic dehydration or hypovolemia, poor fluid or nutritional intake, or a recent clinically significant infection, as per the investigator's judgment.
12. Cancer diagnosis in the past 2 years excluding select skin conditions considered to be fully treated (basal cell or squamous cell carcinomas of the skin) or early-stage cancer with excellent prognosis (eg, some prostate cancer conditions) according to the investigator's judgment.
13. Renal disease (estimated glomerular filtration rate <30 ml/min/1.73m2) based on the investigator's assessment and historical data.
14. Uncontrolled hypertension (systolic blood pressure >160 mm Hg, and/or diastolic blood pressure >100 mm Hg).
15. Significant and uncontrolled thyroid disease according to the investigator's judgment.
16. Any surgery or procedure requiring general anesthesia ≥3 hours, planned, or in the previous 3 months.
17. Poorly regulated type 2 diabetes (HbA1c >9.0%), or type 2 diabetes that is currently treated with insulin, glucagon-like peptide-1 receptor analog (GLP-1 RA), or a sodium-glucose cotransporter-2 (SGLT-2) inhibitor, or type 1 diabetes.
18. Vitamin B12 deficiency per the investigator's judgment, or current use of B-vitamin supplementation >200% daily recommended value according to national standards.
19. Very high or severe hypertriglyceridemia (≥886 mg/dL or 10.0 mmol/L).
20. Participants who are unable to comply with protocol procedures in the opinion of the investigator (if an individual develops a major neurocognitive disorder during the course of the trial, the appropriateness for the individual to continue will be based on the investigator's judgment).
21. Have a personal or hierarchical link with the research team members.
22. Participant who is a shift worker that involves night shifts.
23. Ongoing/planned pregnancy or breastfeeding at screening (female participants who have a positive pregnancy test result before receiving nutritional formulation will be excluded).
24. Participants who follow a ketogenic diet or other diet that is intended to influence ketone levels (eg, prolonged fasting, intermittent fasting, ketogenic meal replacement product regimens), or take ketone-, kMCT-, or coconut oil supplementation, or adhere to a diet that excludes milk product use (eg, vegan diet).
25. Cow's milk protein allergy or intolerance, or other allergy or intolerance to any of the ingredients of the nutritional formulation (eg, medium chain acyl-CoA deficiency, or other fatty acid oxidation disorders).

US protocol specificities:

4. Have MCI (with a clinical phenotype compatible with AD, insidious SVD [ie, no post-stroke cognitive impairment], or mixed AD/SVD) according to the participating site or referring center, as aligned with the National Institute on Aging and the Alzheimer's Association or Mayo Clinic standards for MCI, and additionally informed by a minimum of one of the following objective criteria as assessed by components of the Consortium to Establish a Registry for Alzheimer's Disease neuropsychological battery (CERADNB):

1. Word list memory task: ≤19,
2. Word list recall: ≤5,
3. Fifteen-item subset of the Boston Naming Test (BNT): ≤13,
4. Constructional praxis recall: ≤7, or
5. Total CERAD score: ≤70.

   6. Participants must have an available trial informant willing to attend the following 4 clinic visits with the participant: screening, V1/randomization, V3/12-month visit, and V4/18-month visit.

   9. CDR global score of 0 at screening.

   10. Sexually active females of childbearing potential must practice highly effective methods of contraception with their heterosexual partner (defined in further detail in Appendix 1 of the protocol) or remain abstinent during the trial and for 30 days after the last dose of nutritional formulation. If employing contraception, the highly effective methods of contraception detailed in Appendix 1 of the protocol must be followed.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Preclinical Alzheimer's Cognitive Composite (PACC) score | 12 months
  The change from baseline on the PACC composite cognitive score of episodic memory, timed executive function, and global cognition
  PACC has 4 components:
  * Free and Cued Selective Reminding Test (0 (worst)-96 (best recall);
  * Logical Memory Ib (Immediate Recall) from the WMS-IV (Range 0 (worst)-25 (best recall);
  * Wechsler Adult Intelligence scale - revised: Digit Symbol Substitution Test (DSST): (ranges 0 [none]-93 [best performance])
  * Mini Mental State Examination (Range 0 [worst] - 30 [best performance]).
  Component scores are transformed using an established normalization method into z-scores. Each of 4 component change scores is divided by baseline sample standard deviation (SD) of that component. These z scores are summed to form the composite score. A z-score of 0 is equal to the mean and implies how many SD higher or lower score as compared with baseline score, with increase signifying improvement.

SECONDARY OUTCOMES:
Preclinical Alzheimer's Cognitive Composite (PACC) (components effects) | 12 months
  Individual interventional effects on change from baseline in the individual components of the PACC test (cognitive domains of executive function, episodic memory, and global cognitive function)
  PACC has 4 components:
  * Free and Cued Selective Reminding Test (0 (worst)-96 (best recall);
  * Logical Memory Ib (Immediate Recall) from the WMS-IV (Range 0 (worst)-25 (best recall);
  * Wechsler Adult Intelligence scale - revised: Digit Symbol Substitution Test (DSST): (ranges 0 [none]-93 [best performance])
  * Mini Mental State Examination (Range 0 [worst] - 30 [best performance]).
Montreal Cognitive Assessment (MoCA) score | 12 months
  The change from baseline in the Montreal Cognitive Assessment (MoCA) total score Scale range 0 to 30 - higher score indicates better performance
Preclinical Alzheimer's Cognitive Composite (PACC) accelerated decline | 12 months
  Percentage of participants achieving accelerated cognitive decline, defined as a change from baseline in the PACC z-score of at least 1 SD below the mean
  PACC has 4 components:
  * Free and Cued Selective Reminding Test (0 (worst)-96 (best recall);
  * Logical Memory Ib (Immediate Recall) from the WMS-IV (Range 0 (worst)-25 (best recall);
  * Wechsler Adult Intelligence scale - revised: Digit Symbol Substitution Test (DSST): (ranges 0 [none]-93 [best performance])
  * Mini Mental State Examination (Range 0 [worst] - 30 [best performance]).
  Component scores are transformed using an established normalization method into z-scores. Each of 4 component change scores is divided by baseline sample standard deviation (SD) of that component. These z scores are summed to form the composite score. A z-score of 0 is equal to the mean and implies how many SD higher or lower score as compared with baseline score, with increase signifying improvement.
Wechsler Memory Scale - Fourth Edition (WMS-IV) Logical Memory IIb Delayed Recall Score accelerated decline | 12 months
  Percentage of participants achieving accelerated memory decline, defined as a change from baseline in episodic memory (>3 points) as assessed by the "WMS-IV Logical Memory IIb Delayed Recall Score"
  Wechsler Adult Intelligence scale: Digit Symbol Substitution Test (DSST): (ranges 0 [none]-91 [best performance])
Mini-Mental State Examination (MMSE) score accelerated decline | 12 months
  Percentage of participants achieving accelerated cognitive decline, defined as a change from baseline in the Mini-Mental State Examination (MMSE) total score of <24 or a decline of >3 points Scale range 0 to 30 - higher score indicates better performance
Emergent Adverse Events (Safety and tolerability) | 12 months
  Adverse events (AEs), including gastrointestinal tolerability and nausea, vital signs, changes in blood biomarkers (hematology, liver, kidney) over the course of the trial

CONTACTS AND LOCATIONS:
Locations (30):
- United States (2):
  - Stein Gerontological Institute Inc, Miami, Florida
  - University of Rochester, Rochester, New York
- France (4):
  - Hôpital Pierre Wertheimer, Bron
  - CHU de Montpellier - Hôpital Gui de Chauliac, Montpellier
  - CHU de Nantes - Hôpital Nord Laennec, Nantes
  - CHU de Toulouse - Gerontopole, Toulouse
- Germany (4):
  - Klinikum Bayreuth GmbH - Klinik Hohe Warte, Bayreuth
  - Studienzentrum für Neurologie und Psychiatrie, Böblingen
  - Neuro Centrum Science GmbH, Erbach im Odenwald
  - Universitaetsmedizin Ulm, Ulm
- Italy (8):
  - Foundation Institute G.Giglio, Cefalù
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Azienda Ospedaliera Universitaria Policlinico "Paolo Giaccone", Palermo
  - AOU Policlinico Umberto I - Sapienza Università di Roma, Roma
  - Azienda Ospedaliera SantAndrea, Roma
  - Laboratory of Neuropsyichiatry, Fondazione Santa Lucia IRCCS, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - AO Card. G. Panico, Tricase
- Spain (7):
  - Hospital Universitario del Vinalopó, Alicante
  - Fundaciò ACE, Barcelona
  - HGU Gregorio Marañón, Madrid
  - Unidad de Investigación Neurociencias Centro de Salud San Juan, Salamanca
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès
  - Hospital Universitario Victoria Eugenia, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Switzerland (3):
  - Universitare Altersmedizin FELIX PLATTER, Basel
  - Spitalzentrum Centre Hospitalier Biel-Bienne AG (SZB), Biel
  - CHUV, Lausanne
- United Kingdom (2):
  - Sussex Partnership NHS foundation Trust, Crowborough
  - Hampshire & Isle of Wight Healthcare NHS Foundation Trust, Southampton